CLINICAL TRIAL: NCT04358302
Title: Individual Patient Exposure and Response in Pediatric Lupus
Acronym: iPERSONAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00104621
Record Dates: First submitted 2020-04-16; First posted 2020-04-24 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Systemic Lupus Erythematosus
Keywords: hydroxychloroquine; virtual trial
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Intervention Model Description: Open-label, direct-to-family, adherence and exposure-response study of hydroxychloroquine (HCQ) self-administration in pediatric lupus participants with the use of an electronic pill bottle cap that provides automatic dosing reminders
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Device use (Experimental): All participants will be provided with the electronic pill bottle cap called "Pillsy" to use with their regular HCQ prescription bottles at the start of the study.
  Interventions: Behavioral: Pillsy

INTERVENTIONS:
Behavioral: Pillsy — The electronic pill bottle cap, Pillsy, and its accompanying software application provides reminders to take a scheduled dosage of medication via bottle cap alerts and smartphone push notifications, text messages, and/or automated phone calls. The Pillsy application records dosing dispense date and time when the user opens the bottle. During the first 2 weeks of the trial, the electronic notifications will be disabled to determine a baseline measure of adherence. Within 1 day after Visit 2, the electronic notifications will be turned on for all participants, resulting in a series of alerts (via electronic pill bottle cap alerts and smartphone push notifications, text message, and/or automated phone calls).
  The electronic pill bottle cap, Pillsy, is a commercially available device marketed to consumers. The electronic pill bottle cap does not capture or store PHI. Quick tips on how to use Pillsy can be found at https://www.pillsy.com/instructions

SUMMARY:
The purpose of this research study is to see if an electronic pill bottle cap can help children and teens with systemic lupus better remember to take their medicine. It will also gather information on the best dose of hydroxychloroquine (Plaquenil®) for children and teens. Participants in this study will continue to take their usual medication as prescribed by their doctors. Participants will receive an electronic pill bottle cap, a smartphone, and a Fitbit. Over 6 months, a nurse will visit each participant 4 times to ask questions about symptoms, draw blood, and take a urine sample. After the study, participants will be able to keep the electronic pill bottle cap and Fitbit, but will return the smartphone.

DETAILED DESCRIPTION:
This is an exploratory Phase 2, single site, open-label, direct-to-family, adherence and exposure-response study of hydroxychloroquine (HCQ) in pediatric systemic lupus. The study will measure a participant's adherence to HCQ self-administration using an electronic pill bottle cap that records date/time of bottle opening and provides participants with a reminder when a dosage is due and/or missed. All participants will be provided with the electronic pill bottle cap to use with their regular HCQ prescription at the start of the study. For the first 2 weeks of the trial, the electronic notifications will be disabled to determine a baseline measure of adherence. Within 1 day after Visit 2, the electronic notifications will be turned on for all participants, resulting in a series of alerts (via electronic pill bottle cap alerts and smartphone push notifications, text message, and/or automated phone calls). Participants will continue to receive notifications via the electronic pill bottle cap through Visit 4. Throughout the study, participants will undergo a series of blood draws and urinalysis collections, and be asked to complete various questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent form and assent, when necessary
2. Age 5-17.5 years at consent
3. Enrolled in the CARRA Registry with a diagnosis of systemic lupus erythematosus as documented in the CARRA Registry
4. Receiving hydroxychloroquine as standard of care for ≥ 3 months
5. Participant and Caregiver primary language of English
6. Willing and able to comply with study procedures, at the discretion of the study principal investigator
7. Access to internet

Exclusion Criteria:

There are no pre-defined exclusion criterion for this trial.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2021-06-16 (Actual); Study Completion 2021-06-16 (Actual)

PRIMARY OUTCOMES:
Change in proportion of dispensed doses from the first two weeks (baseline) to last two weeks of study (device use) | Days 1-14 compared to days 166-180 (+/- 30)
  The Pillsy device will record the number of dispensed doses

SECONDARY OUTCOMES:
Adherence to hydroxychloroquine using the Medication Adherence Self-Reported Inventory (MASRI) score | Up to 6 months
  The MASRI is a concise, self-administered survey completed by the patient at study visits. The MASRI is a patient-reported numeric estimate of medication adherence rate (0-100%) with non-adherence defined as MASRI <80% and adherence defined as >/=80%.
Adherence to hydroxychloroquine using plasma drug levels | Up to 6 months
  Plasma drug levels will be measured by patient blood collection at study visits
Adherence to hydroxychloroquine using electronic pill counts | Up to 6 months
  Electronic pill counts will be obtained by the Pillsy device
Adherence to hydroxychloroquine using manual pill counts | Up to 6 months
  Manual pill counts will be conducted by the nurse at study visits
Disease activity as measured by Systemic Lupus Activity Questionnaire (SLAQ) score | Up to 6 months
  The SLAQ is a concise, self-administered survey completed by the patient at study visits. The SLAQ measures patient-reported disease activity and scores range from 0-44, with 0 representing no disease activity and 44 representing maximum disease activity.
Disease activity as measured by the Systemic Lupus Erythematosus Disease Activity Index (SLEDAI-2K) score collected through a remote teleresearch exam | Up to 2 months
  A physician will conduct a remote SLEDAI-2K assessment of the patient at study visit 1. The SLEDAI-2K measures physician-reported disease activity and scores range from 0-105, with 0 representing no disease activity and 105 representing maximum disease activity. A score of >/=6 represents clinically important disease activity and a reduction of at least 4 represents clinically meaningful improvement in disease activity.
Disease activity as measured by the Systemic Lupus Erythematosus Disease Activity Index (SLEDAI-2K) score recorded in the CARRA Registry | Up to 6 months
  SLEDAI-2K score recorded from the patient's closest CARRA Registry visit relative to visit 1

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Balevic, MD, MHS, Principal Investigator — Duke Clinical Research Institute
Locations (1):
- Duke Clinical Research Institute, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Balevic SJ, Randell R, Weiner D, Beard C, Schanberg LE, Hornik CP, Cohen-Wolkowiez M, Gonzalez D; with the CARRA Registry investigators. Pharmacokinetics of hydroxychloroquine in paediatric lupus: data from a novel, direct-to-family clinical trial. Lupus Sci Med. 2022 Nov;9(1):e000811. doi: 10.1136/lupus-2022-000811. PMID 36328395
- [Derived] Randell RL, Singler L, Cunningham A, Schanberg LE, Cohen-Wolkowiez M, Hornik CP, Balevic SJ; with the CARRA Registry investigators. Delivering clinical trials at home: protocol, design and implementation of a direct-to-family paediatric lupus trial. Lupus Sci Med. 2021 May;8(1):e000494. doi: 10.1136/lupus-2021-000494. PMID 33963084